CLINICAL TRIAL: NCT01549015
Title: Open, Prospective, Diagnostic, Multicentre Study in Healthy Subjects, Patients With Urea Cycle Disorders (UCD), and Carriers of UCD Mutations, to Evaluate in Vivo Ureagenesis Measured After a Single Application of Sodium [1,2-13C]-Acetate
Brief Title: Study in Healthy Subjects, Patients With Urea Cycle Disorders (UCD) and Carriers of UCD Mutations to Evaluate Urea Cycle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cytonet GmbH & Co. KG (Industry)
Collaborators: CRS Clinical Research Services Mannheim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCD09; 2011-002472-16 (EudraCT Number)
Record Dates: First submitted 2012-01-16; First posted 2012-03-08 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Urea Cycle Disorders
Keywords: Urea Cycle Defects; CPSD; OTCD; ASSD; ASLD
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: oral administration of Sodium [1,2-13C]-Acetate — single dose of 0.55 mg/kg 13C-Acetate given orally of via a naso-gastric tube

SUMMARY:
This diagnostic study will be performed to investigate the performance of the urea cycle in healthy subjects, asymptomatic carriers of Urea Cycle Disorders (UCD) mutations and subjects with genetically proven urea cycle disorders. The ureagenesis rate will be measured by 13C incorporation assay, a method for in vivo measurement of urea cycle performance with stable isotopes.

DETAILED DESCRIPTION:
In this diagnostic study CCD09, the urea metabolism in UCD subjects (patients and carriers) and healthy subjects of different age and sex will be assessed by measurement of the incorporation of 13C from orally taken sodium [1,2-13C]-acetate into urea by 13C stable isotope ratio detection. The aim of the study is to determine the 13C urea production and to quantify the total urea production in healthy subject, gene defect carrier or patient as marker for the functioning of the urea cycle. Since there are still only few data available using this specific method for measurement of urea cycle performance, the aim of this study CCD09 is to gain additional results on the 13C assay. To this end, comparison will be made between 13C urea production observed in healthy subjects, UCD patients, and asymptomatic mutation carriers.

An evaluation of this study may also enable the treating physician to better judge the severity of disease and the future risk of metabolic decompensations in patients as well as the potential risk for so far asymptomatic carriers.

ELIGIBILITY:
Inclusion Criteria:

All study groups:

• Written informed consent given by subjects or his/her parents/legal guardians who are able to understand and follow instructions related to the study

Group 1 Healthy Volunteers:

* Age: 18 - 65 years
* Healthy subjects
* No clinical or laboratory parameter outside normal ranges at screening and judged as clinically relevant by the investigator

Group 2 Symptomatic UCD patients with genetically confirmed CPSD, OTCD, ASSD, or ASLD:

Age: 0 - 65 years

* Symptomatic subjects with genetically confirmed Carbamylphosphate synthetase I Deficiency [CPSD], Ornithine Transcarbamylase Deficiency [OTCD], Argininosuccinate Synthetase Deficiency [Citrullinaemia type I], Argininosuccinate Lyase Deficiency [ASLD]
* at least 1 metabolic decompensation with clinical signs of hyperammonemia in medical history or genetically confirmed and prospectively treated siblings of symptomatic patients, even without clinical symptoms
* Confirmed diagnosis and medical history available (in particular number and severity of metabolic crises)

Group 3 Asymptomatic carriers of UCD mutations:

* Age: 0 - 65 years
* Asymptomatic carriers of mutations for Carbamylphosphate synthetase I Deficiency [CPSD], Ornithine Transcarbamylase Deficiency [OTCD], Argininosuccinate Synthetase Deficiency [Citrullinaemia type 1], Argininosuccinate Lyase Deficiency [ASLD] no dietary protein restriction, no intake of ammonia scavenging drugs, no known metabolic decompensation with clinical signs of hyperammonemia

Group 4:

* Infants between 8 - 10 kg body weight Symptomatic subjects with genetically confirmed Carbamylphosphate synthetase I Deficiency [CPSD] Ornithine Transcarbamylase Deficiency [OTCD] Argininosuccinate Synthetase Deficiency [Citrullinaemia type I] Argininosuccinate Lyase Deficiency [ASLD] at least 1 metabolic decompensation with clinical signs of hyperammonemia in medical history or genetically confirmed and prospectively treated siblings of symptomatic patients, even without clinical symptoms
* Confirmed diagnosis and medical history available (in particular number and severity of metabolic crises

Exclusion Criteria:

* Acute illness, including vomiting, fever or other sign of infection
* Participation in other invasive clinical trials within 30 days prior to inclusion
* Liver or renal disease
* Acute seizures
* Coma
* Bleeding disorder
* Blood ammonia > 100 µmol/l for patients with a urea cycle disorder and blood ammonia > normal for healthy probands and asymptomatic carriers
* Metabolic acidosis
* Pregnancy or lactation
* Body weight < 8kg
* Chronic somatic or psychiatric disease not related to UCD

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Formation of 13C-urea in plasma | 0 - 240 Minutes

SECONDARY OUTCOMES:
Vital signs | 0-240 min
  blood pressure, heart rate, temperature and respiratory rate at enrollment and after completion
Complete blood count without differential | at enrollement
Adverse events | 0-240 mins
Ammonia, Amino acids, Urea in serum | 0-240 min
CRP | at enrollment
Venous lactate and blood gases: pH, pCO2, pO2, bicarbonate | at enrollment
Blood glucose | 0 - 240 min
pH and bicarbonate | 20 and 60 mins after administration

CONTACTS AND LOCATIONS:
Overall Officials: Georg F Hoffmann, Prof Dr med, Principal Investigator — Universitätsklinikum Heidelberg Klinik für Kinderheilkunde I
Locations (4):
- Germany (4):
  - CRS Clinical Research Services GmbH (Phase I Unit), Mönchengladbach
  - Medizinische Hochschule Hannover, Klinik für Kinderheilkunde, Hanover
  - Universitätsklinikum Heidelberg Klinik für Kinderheilkunde I, Heidelberg
  - Universitätsklinikum Münster, Zentrum für Kinder- und Jugendmedizin, Münster